CLINICAL TRIAL: NCT03899064
Title: A 6-Week, Randomized Study to Evaluate the Potential of MC2-01 Cream to Induce Photoallergic Skin Reaction in Healthy Subjects, Using a Controlled Photopatch Test Design
Brief Title: Evaluation of Potential Development of Photoallergic Skin Reaction After Use of MC2-01 Cream
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MC2 Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MC2-01-C10
Record Dates: First submitted 2019-03-20; First posted 2019-04-02 (Actual); Results first posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-02

CONDITIONS: Photoallergy
MeSH Terms: conditions — Dermatitis, Photoallergic | interventions — Radiation

STUDY DESIGN:
Intervention Model Description: The study consist of an Induction phase, where treatments (MC2-01 Cream, MC2-01 vehicle) were applied to 2 test sites each (n=4), followed by irradiation/non-irradiation and evaluation 24, 48 or 72 hours post-irradiation. This was repeated in total 6 times over an 3 weeks period. The induction phase was followed by a challenge phase, where treatments (MC2-01 Cream, MC2-01 vehicle) were applied to each two naive test sites and another naive test site was untreated. 24 hours of product application, one of each test sites (MC2-01 Cream, MC2-01 vehicle) + the untreated test site were irradiated. Possible changes in dermal reaction (erythema and edema) was evaluated at all 5 test sites, 24, 48 and 72 hours post-irradiation.
Who Masked: Participant, Outcomes Assessor
Masking Description: The tests sites (M2-01 Cream, MC2-01 vehicle, control) will not be blinded to the site staff involved in the preparation/application and removal of treatments. The subjects and the trained assessor will be blinded to the IPs and treatment allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Induction:MC2-01 Cream, irradiation (Experimental): Applications with MC2-01 Cream (calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%), followed by irradiation
  Interventions: Drug: Induction: Application of MC2-01 Cream, irradiation
- Induction: MC2-01 Cream, no irradiation (Experimental): Applications with MC2-01 Cream (calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%), no irradiation
  Interventions: Drug: Induction: Application of MC2-01 Cream, no irradiation
- Induction: MC2-01 vehicle, irradiation (Experimental): Applications with MC2-01 vehicle, followed by irradiation
  Interventions: Drug: Induction: Applications of MC2-01 vehicle, irradiation
- Induction: MC2-01 vehicle, no irradiation (Experimental): Applications with MC2-01 vehicle, no irradiation
  Interventions: Drug: Induction: Applications of MC2-01 vehicle, no irradiation
- Challenge: MC2-01 Cream, irradiation (Experimental): Application with MC2-01 Cream (calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%), followed by irradiation
  Interventions: Drug: Challenge: Application of MC2-01 Cream, irradiation
- Challenge: MC2-01 Cream, No irradiation (Experimental): Application with MC2-01 Cream (calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%), no irradiation
  Interventions: Drug: Challenge: Application of MC2-01 Cream, no irradiation
- Challenge: MC2-01 vehicle, irradiation (Experimental): Application with MC2-01 vehicle, followed by irradiation
  Interventions: Drug: Challenge: Applications of MC2-01 vehicle, irradiation
- Challenge: MC2-01 vehicle, no irradiation (Experimental): Application with MC2-01 vehicle, no irradiation
  Interventions: Drug: Challenge: Applications of MC2-01 vehicle, no irradiation
- Challenge: Control, irradiation (Experimental): No application, but irradiation
  Interventions: Drug: Challenge: Control, irradiation

INTERVENTIONS:
Drug: Induction: Application of MC2-01 Cream, irradiation — Repeated applications of MC2-01 Cream (CAL/BDP, 0.005%/0.064%), followed by irradiation. Visual evaluation of application site using a visual scale that rated the degree of erythema, edema and other signs of cutaneous irritation
  Arms: Induction:MC2-01 Cream, irradiation
Drug: Induction: Application of MC2-01 Cream, no irradiation — Repeated applications of MC2-01 Cream, CAL/BDP, 0.005%/0.064%, no irradiation. Visual evaluation of application site using a visual scale that rated the degree of erythema, edema and other signs of cutaneous irritation
  Arms: Induction: MC2-01 Cream, no irradiation
Drug: Induction: Applications of MC2-01 vehicle, irradiation — Repeated applications of MC2-01 cream, followed by irradiation. Visual evaluation of application site using a visual scale that rated the degree of erythema, edema and other signs of cutaneous irritation
  Arms: Induction: MC2-01 vehicle, irradiation
Drug: Induction: Applications of MC2-01 vehicle, no irradiation — Repeated applications of MC2-01 vehicle, no irradiation. Visual evaluation of application site using a visual scale that rated the degree of erythema, edema and other signs of cutaneous irritation
  Arms: Induction: MC2-01 vehicle, no irradiation
Drug: Challenge: Application of MC2-01 Cream, irradiation — Single application of MC2-01 Cream (CAL/BDP, 0.005%/0.064%), followed by irradiation. Visual evaluation of application site using a visual scale that rated the degree of erythema and edema
  Arms: Challenge: MC2-01 Cream, irradiation
Drug: Challenge: Application of MC2-01 Cream, no irradiation — Single application of MC2-01 Cream (CAL/BDP, 0.005%/0.064%), no irradiation. Visual evaluation of application site using a visual scale that rated the degree of erythema and edema
  Arms: Challenge: MC2-01 Cream, No irradiation
Drug: Challenge: Applications of MC2-01 vehicle, irradiation — Single application of MC2-01 vehicle, followed by irradiation. Visual evaluation of application site using a visual scale that rated the degree of erythema and edema
  Arms: Challenge: MC2-01 vehicle, irradiation
Drug: Challenge: Applications of MC2-01 vehicle, no irradiation — Single application of MC2-01 vehicle, no irradiation. Visual evaluation of application site using a visual scale that rated the degree of erythema and edema
  Arms: Challenge: MC2-01 vehicle, no irradiation
Drug: Challenge: Control, irradiation — No application, but irradiation. Visual evaluation of application site using a visual scale that rated the degree of erythema and edema
  Arms: Challenge: Control, irradiation

SUMMARY:
This trial is a 6-week, Randomized study evaluating the potential of MC2-01 Cream to induce a photoallergic skin reaction in Healthy subjects, using a controlled photopatch test design.

DETAILED DESCRIPTION:
The study evaluates the potential of MC2-01(CAL/BDP 0.005/0.064 w/w%) Cream to induce a photoallergic skin reaction. Because MC2-01 Cream is formulated for topical use and has shown to absorb light within the range of natural sunlight, it is necessary to determine the potential of this product to cause a photoallergic reaction after application to the skin.

ELIGIBILITY:
Inclusion Criteria:

* Is a healthy male or female
* Is 18 years of age or older
* Agree not to participate in any clinical or patch test studies at Day 1 through study completion
* Females or childbearing potential must use a highly effective method of contraception for one month prior to Screening and until the end of study visit has been performed
* In the case of a female of childbearing potential, has a negative urine pregnancy test on Day 1 prior to randomization and are willing to submit to a urine pregnancy test at the end of study
* In the case of a female of childbearing potential, has had a hysterectomy or is postmenopausal
* Is free of any systemic or dermatological disorder, which, in the opinion of the Investigator, will interfere with the study results or increase the risk of AEs.
* Has uniformly-colored skin on the intrascapular region of the back which will allow discernment of erythema, and has Fitzpatrick skin types I, II or III
* Complete a medical screening procedure
* Read, understand and sign an informed consent

Exclusion Criteria:

* Has a history of photosensitivity or photoallergy
* Has any visible skin disease at the application site which, in the opinion of the Investigator, will interfere with the evaluation of the test site reaction
* Current or past history of hypercalcemia, vitamin D toxicity, severe renal insufficiency or severe hepatic disorders
* Is using systemic/topical corticosteroids within 3 weeks prior to and/or during the study or systemic/topical antihistamines 72 hours prior to and during the study
* Is not willing to refrain from using systemic/topical anti-inflammatory analgesics (81 mg aspirin and occasional use of acetaminophen will be permitted)
* Are taking medication known to cause phototoxic reaction
* Is using medication which, in the opinion of the Investigator, will interfere with the study results
* Is unwilling or unable to refrain from the use of sunscreens, cosmetics, creams, ointments, lotions or similar products on the back during the study
* Has psoriasis and/or atopic dermatitis/eczema
* Has a known sensitivity or allergy to constituents of the materials being evaluated
* Is a female who is pregnant, plans to become pregnant during the study, or is breast feeding a child
* Has damaged skin in or around the test sites, including sunburn, excessively deep tans, uneven skin tones, tattoos, scars excessive hair, numerous freckles or other disfigurations of the test site
* Has received treatment for any type of internal cancer within 5 years prior to study entry
* Has a history of, or are currently being treated for skin cancer and/or hepatitis
* Has a history or, or is currently being treated for diabetes
* Has any condition that might compromise study results
* Is expected to sunbathe or use tanning salons during the study
* Has a history of adverse response to UV-sun lamps/sunlight exposure
* Is currently participating in any clinical testing
* Has any known sensitivity to adhesives
* Has received any investigational drug(s) within 28 days from Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S Dosik, MD, Principal Investigator — TKL Research
Locations (1):
- TKL Research Inc., Fair Lawn, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Single site study

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject First Visit: 18-Feb-2019; Last Subject Last Visit: 05-Apr-2019
Pre-assignment Details: This study was a randomized, double-blind, controlled, within-subject comparison study to evaluate the potential of MC2-01 cream to induce a photoallergic skin reaction.
  The study consist of a 3-week Induction phase, followed by a Challenge phase.
Groups:
- Test Sites: 5 test sites on the subject's back defined as:
  1. Applications with MC2-01 Cream (calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%), followed by irradiation
  2. Application with MC2-01 Cream (calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%), no irradiation
  3. Applications with MC2-01 vehicle, followed by irradiation
  4. Applications with MC2-01 vehicle, no irradiation
  5. No application, but irradiation
Period: Overall Study
Arm/Group | Test Sites
Started | 58
MC2-01 Cream, Irradiation | 58
MC2-01 Cream, No Irradiation | 58
MC2-01 Vehicle, Irradiation | 58
MC2-01 Vehicle, no Irradiation | 58
Control, Irradiation | 58
Completed | 51
Not Completed | 7
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 2
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Arm/Group | Test Sites
Number analyzed (Participants) | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (11.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 56
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 58
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Measure Description: Fitzpatrick Skin Type is a method to describe the individual skin types in the following 6 categories:
  I - Pale white skin, blue/hazel eyes, blond/red hair; II - Fair skin, blue eyes III - Darker white skin; IV - Light brown skin; V - Brown skin; VI - Dark brown or black skin
  Participants
    I | 2
    II | 18
    III | 38
    IV | 0
    V | 0
    VI | 0

OUTCOME MEASURES:

1. Primary Outcome: Within-subject Comparison of Dermal Reaction by the Overall Numeric Rating of Erythema and Edema at 5 Defined Test Sites, After Application of MC2-01 Cream, MC2-01 Vehicle or Untreated at Defined Test Sites, Followed by Irradiation.
Description: After an induction phase, where subjects were treated with MC2-01 Cream, MC2-01 vehicle and irradiation, the challenge phase was initiated.
  MC2-01 Cream and MC2-01 vehicle was applied to each two naive test sites. Another naive test site was untreated. 24 hours after product application, one of each test site (MC2-01 Cream, MC2-01 vehicle) + the untreated site were irradiated. Possible changes in dermal reaction (erythema and edema) was evaluated at all 5 test sites 24, 48 and 72 hours post-irradiation and these evaluations are the outcome measure of the study.
  The following visual scores was used to express the response observed at each timepoints: Erythema: 0-3 where 0 represents no reaction and 3 represents marked/severe erythema. Edema: 0-2 where 0 represents no reaction and 2 represents definite edema with erosion/vesiculation. The diagnosis of photosensitization response will be made by the investigator based on review of the scored skin responses of both erythema and edema.
Time Frame: 24 hours
Population: As the study is a within subject evaluation of dermal reactions, after application on two sites with MC2-01 cream, two sites with MC2-01 vehicle and one site untreated, followed by either irradiation or non-irradiation, all subjects received all 5 different treatments.
Measure: Count of Participants; unit: Participants
Arm/Group | Test Sites
Number analyzed (Participants) | 51
Participants
  MC2-01 Cream, irradiation: No erythema/edema | 48
  MC2-01 Cream, irradiation: Mild, definite erythema/edema | 3
  MC2-01 Cream, irradiation: Moderate erythema/defined edema | 0
  MC2-01 Cream, irradiation: Marked/severe erythema | 0
  MC2-01 Cream, No irradiation: No erythema/edema | 49
  MC2-01 Cream, No irradiation: Mild, definite erythema/edema | 2
  MC2-01 Cream, No irradiation: Moderate erythema/defined edema | 0
  MC2-01 Cream, No irradiation: Marked/severe erythema | 0
  MC2-01 vehicle, irradiation: No erythema/edema | 49
  MC2-01 vehicle, irradiation: Mild, definite erythema/edema | 2
  MC2-01 vehicle, irradiation: Moderate erythema/defined edema | 0
  MC2-01 vehicle, irradiation: Marked/severe erythema | 0
  MC2-01 vehicle, no irradiation: No erythema/edema | 50
  MC2-01 vehicle, no irradiation: Mild, definite erythema/edema | 1
  MC2-01 vehicle, no irradiation: Moderate erythema/defined edema | 0
  MC2-01 vehicle, no irradiation: Marked/severe erythema | 0
  Control, Irradiation: No erythema/edema | 47
  Control, Irradiation: Mild, definite erythema/edema | 4
  Control, Irradiation: Moderate erythema/defined edema | 0
  Control, Irradiation: Marked/severe erythema | 0

2. Primary Outcome: Within-subject Comparison of Dermal Reaction by the Overall Numeric Rating of Erythema and Edema at 5 Defined Test Sites, After Application of MC2-01 Cream, MC2-01 Vehicle or Untreated at Defined Test Sites, Followed by Irradiation.
Description: After an induction phase, where subjects were treated with MC2-01 Cream, MC2-01 vehicle and irradiation, the challenge phase was initiated.
  MC2-01 Cream and MC2-01 vehicle was applied to each two naive test sites. Another two naive test sites were untreated. 24 hours of product application, one of each test site (MC2-01 Cream, MC2-01 vehicle and untreated) were irradiated.
  Possible changes in dermal reaction (erythema and edema) was evaluated at all 6 test sites, 24, 48 and 72 hours post-irradiation and these evaluations are the outcome measure of the study. The following visual scores was used to express the response observed at each timepoints: Erythema: 0-3 where 0 represents no reaction and 3 represents marked/severe erythema. Edema: 0-2 where 0 represents no reaction and 2 represents definite edema with erosion/vesiculation. The diagnosis of photosensitization response will be made by the investigator based on review of the scored skin responses of both erythema and edema.
Time Frame: 48 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Test Sites
Number analyzed (Participants) | 51
Participants
  MC2-01 Cream, irradiation: No erythema/edema | 48
  MC2-01 Cream, irradiation: Mild, definite erythema/edema | 3
  MC2-01 Cream, irradiation: Moderate erythema/defined edema | 0
  MC2-01 Cream, irradiation: Marked/severe erythema | 0
  MC2-01 Cream, No irradiation: No erythema/edema | 51
  MC2-01 Cream, No irradiation: Mild, definite erythema/edema | 0
  MC2-01 Cream, No irradiation: Moderate erythema/defined edema | 0
  MC2-01 Cream, No irradiation: Marked/severe erythema | 0
  MC2-01 vehicle, irradiation: No erythema/edema | 48
  MC2-01 vehicle, irradiation: Mild, definite erythema/edema | 3
  MC2-01 vehicle, irradiation: Moderate erythema/defined edema | 0
  MC2-01 vehicle, irradiation: Marked/severe erythema | 0
  MC2-01 vehicle, no irradiation: No erythema/edema | 50
  MC2-01 vehicle, no irradiation: Mild, definite erythema/edema | 1
  MC2-01 vehicle, no irradiation: Moderate erythema/defined edema | 0
  MC2-01 vehicle, no irradiation: Marked/severe erythema | 0
  Control, Irradiation: No erythema/edema | 48
  Control, Irradiation: Mild, definite erythema/edema | 3
  Control, Irradiation: Moderate erythema/defined edema | 0
  Control, Irradiation: Marked/severe erythema | 0

3. Primary Outcome: Within-subject Comparison of Dermal Reaction by the Overall Numeric Rating of Erythema and Edema at 5 Defined Test Sites, After Application of MC2-01 Cream, MC2-01 Vehicle or Untreated at Defined Test Sites, Followed by Irradiation.
Description: as for outcome 2
Time Frame: 72 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Test Sites
Number analyzed (Participants) | 51
Participants
  MC2-01 Cream, irradiation: No erythema/edema | 51
  MC2-01 Cream, irradiation: Mild, definite erythema/edema | 0
  MC2-01 Cream, irradiation: Moderate erythema/defined edema | 0
  MC2-01 Cream, irradiation: Marked/severe erythema | 0
  MC2-01 Cream, No irradiation: No erythema/edema | 51
  MC2-01 Cream, No irradiation: Mild, definite erythema/edema | 0
  MC2-01 Cream, No irradiation: Moderate erythema/defined edema | 0
  MC2-01 Cream, No irradiation: Marked/severe erythema | 0
  MC2-01 vehicle, irradiation: No erythema/edema | 50
  MC2-01 vehicle, irradiation: Mild, definite erythema/edema | 1
  MC2-01 vehicle, irradiation: Moderate erythema/defined edema | 0
  MC2-01 vehicle, irradiation: Marked/severe erythema | 0
  MC2-01 vehicle, no irradiation: No erythema/edema | 51
  MC2-01 vehicle, no irradiation: Mild, definite erythema/edema | 0
  MC2-01 vehicle, no irradiation: Moderate erythema/defined edema | 0
  MC2-01 vehicle, no irradiation: Marked/severe erythema | 0
  Control, Irradiation: No erythema/edema | 51
  Control, Irradiation: Mild, definite erythema/edema | 0
  Control, Irradiation: Moderate erythema/defined edema | 0
  Control, Irradiation: Marked/severe erythema | 0

ADVERSE EVENTS:
Time Frame: AEs were collected/assessed from the time of the informed consent was signed by the subject at the screening visit and during both the induction phase, which consisted of 3 weeks, and the challenge phase, which consisted of 4 days. The 4th day in the challenge phase was considered the last visit for the subjects. AEs assessed as reasonably possibly related to the treatment had to be followed until they were resolved or until the medical condition of the subject was stable.
Description: 58 patients participated in the study and all patients received all 5 types of treatments. Therefore data for the 'All-Cause Mortality', 'Serious Adverse Events' and 'Other Adverse Events' fields are included and assessed for all types of medication.
Arm/Group | Test Sites
All-Cause Mortality (participants affected / at risk) | 0/58
Serious Adverse Events (participants affected / at risk) | 0/58
Other Adverse Events (participants affected / at risk) | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/64/NCT03899064/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-08): https://cdn.clinicaltrials.gov/large-docs/64/NCT03899064/SAP_001.pdf